CLINICAL TRIAL: NCT07067229
Title: Non-invasive Brain Stimulation and Exercise Intervention for Patients With Motor Neuron Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COA No. 1142/2024
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: Amyotrophic Lateral Sclerosis; Transcranial Magnetic Stimulation; Intervention; Augmented Reality
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized intervention group (Experimental): Participants will receive personalised repetitive transcranial magnetic stimulation mixed reality.
  Interventions: Device: Personalized rTMS
- Standard intervention group (Active Comparator): Participants will receive standard repetitive transcranial magnetic stimulation plus mixed reality.
  Interventions: Device: Standard rTMS
- Sham group (Sham Comparator): Participants will receive sham repetitive transcranial magnetic stimulation mixed reality.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Personalized rTMS — Personalized repetitive transcranial magnetic stimulation (TMS) together with mixed-reality (MR) exercise
  Arms: Personalized intervention group
Device: Standard rTMS — Standard repetitive transcranial magnetic stimulation (TMS) together with mixed-reality (MR) exercise
  Arms: Standard intervention group
Device: Sham rTMS — Sham rTMS together with mixed-reality (MR) exercise
  Arms: Sham group

SUMMARY:
Motor neuron disease (MND) is a progressive neurological disorder involving degeneration of motor neurons, leading to muscle weakness, speech and swallowing difficulties, and respiratory failure. This study aims to develop a novel treatment approach combining personalized repetitive transcranial magnetic stimulation (rTMS) with mixed reality (MR) exercise-based games (exergames) to slow disease progression and improve quality of life. In this randomised controlled trial study will compare three groups: (1) rTMS with MR exercise (personalized intervention), (2) rTMS with MR exercise (standard intervention), and (3) sham rTMS with MR exercise. Outcomes will be assessed at baseline, 3 months, and 6 months post intervention. The long-term goal is to implement this approach in clinical settings to enhance care for people with MND.

DETAILED DESCRIPTION:
After screening process, eligible participants will be invited to visit Chula Neuroscience Center for the baseline assessments which will take proximately 2 hours.

The baseline assessments will be as follow:

1. Demographic information such as age, sex, body height, body weight, body mass index, date of diagnosis, type of MND, and current medications.
2. Questionnaires including amyotrophic lateral sclerosis functional rating scale - revised version (ALSFRS-R), penn upper motor neuron score (PUMNS), patient health questionnaire (PHQ-9), and EuroQol 5-Dimension 5-level (EQ-5D-5L).
3. Clinical assessments including hand grip test, pinch grip test, and hand function.
4. Lung function tests such as forced vital capacity (FVC).
5. Neurophysiological assessment by using transcranial magnetic stimulation (TMS)
6. Electromyography (EMG) including compound muscle action potential (CMAP), motor unit number estimation (MScan fit-MUNE), and motor unit number index (MUNIX).
7. Magnetic resonance imaging (MRI)

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 18 and 80 years
* Diagnosed with any type of motor neuron disease (MND)
* Have mild to moderate severity, as assessed by the Sinaki-Mulder scale, with a severity level between 1 and 3

Exclusion Criteria:

* History of other neurological disorders, such as stroke
* Use of ventilatory support
* Severe dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Amyotrophic Lateral Sclerosis Functional rating scale - revised version (ALSFRS-R) | ALSFRS-R will be measured at three time points (baseline, 3-month, and 6-month post intervention).
  The Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) is a 12-item questionnaire used to assess functional ability in people with ALS across four domains: bulbar, fine motor, gross motor, and respiratory function. Each item is scored from 0 (unable) to 4 (normal), with a total score ranging from 0 to 48. It can be self-reported or clinician-administered in person, by phone, or online. Lower scores indicate greater disability. The ALSFRS-R is used to monitor disease progression and guide clinical care.
Muscle evoke potential (MEP) | MEP will be mesured at three time points (baseline, 3-month, and 6-month post intervention).
  Participants will be stimulated at the primary motor cortex by transcranial magnetic stimulation to measure cortical excitability, which sends the motor outputs to Tibialis Anterior (TA) and Abductor Pollicis Brevis (APB) muscles. The MEP will be used to assess muscle activity in these muscles during the stimulation. The MEP will be measured in mV.
Motor unit number estimation (MScan fit-MUNE) | MScan fit-MUNE will be mesured at three time points (baseline, 3-month, and 6-month post intervention).
  For MScan fit-MUNE, CMAP is recorded at multiple stimulation intensities. The MScan fit-MUNE software then generates a curve representing the relationship between stimulation intensity and CMAP amplitude. A mathematical model is fitted to this curve to estimate the number of motor units contributing to the generation of the CMAP.
Motor unit number index (MUNIX) | MUNIX will be measured at three time points (baseline, 3-month, and 6-month post intervention).
  For MUNIX (Motor Unit Number Index), the procedure begins with recording the CMAP. Then, the participant is asked to gently contract the muscle. During this contraction, the interference pattern of muscle electrical activity is recorded. The MUNIX value is calculated by analyzing the ratio between the CMAP amplitude and the amplitude of the interference pattern. This provides an estimate of motor unit function.
Cortical silent period (CSP) | Muscle evoke potential will be measured at three time points (baseline, 3-month, and 6-month post intervention).
  Participants will be stimulated at the primary motor cortex by transcranial magnetic stimulation to measure cortical excitability, which sends the motor outputs to Tibialis Anterior (TA) and Abductor Pollicis Brevis (APB) muscles. The CSP will be used to assess muscle activity in these muscles during the stimulation. The CSP will be measured in ms.

SECONDARY OUTCOMES:
Muscle mass | Muscle mass will be measured at three time points (baseline, 3-month, and 6-month post intervention).
  We will used the bioelectrical impedance analysis (BIA), which is a method used for measuring body composition.Participants will be asked to step on to the BIA device, placing their feet on the foot electrodes. The muscle mass will be recored in kilograms.
Body mass index (BMI) | BMI will be measured at three time point (baseline, 3-month, 6-month post intervention).
  We will used the bioelectrical impedance analysis (BIA), which is a method used for measuring body composition.Participants will be asked to step on to the BIA device, placing their feet on the foot electrodes. The BMI will be recored in kg/m^2.
Hand grip test | Hand grip test will be measured at three time points (baseline, 3-month, and 6-month post intervention).
  The Hand Grip Test is an objective measure of isometric grip strength, commonly used to assess overall muscle strength and functional status. The test is performed using a handheld dynamometer, which the participant squeezes with maximum effort, typically while seated with the elbow at a 90-degree angle. The test is usually repeated three times per hand, and the highest or average value measured in kilograms is recorded. Lower grip strength is associated with reduced physical function and is often used as an indicator of frailty, sarcopenia, or neuromuscular decline.
Pinch grip test | Pinch grip test will be measured at three time points (baseline, 3-month, and 6-month post intervention).
  The Pinch Grip Test is used to assess the strength of the thumb muscles in individuals with motor neuron disease (MND). Participants are asked to hold a pinch grip dynamometer with their arm positioned at a 90-degree angle and squeeze as hard as possible for 3 to 5 seconds. Each set consists of 10 repetitions, and the test includes 5 sets in total, with a 1-minute rest between sets. The goal is to measure the maximum force generated during the test. Afterward, participants are instructed to maintain a pinch force at 50% ± 5% of their maximum strength for as long as possible. Results are recorded in kilograms (kg) and duration (seconds).
Hand function | Hand function will be measured at three time points (baseline, 3-month, and 6-month post intervention).
  Hand function will be assessed using the Wolf Motor Function Test (WMFT) to evaluate gross motor movements, such as placing the hand on a table, placing the arm on a box, and extending the arm. The Jebsen-Taylor Test of Hand Function will be used to assess fine motor movements, such as picking up objects, grasping a can, and handling a paperclip. The outcomes will be recorded as the time taken to complete each task.
Penn upper motor neuron score (PUMNS) | PUMNS will be measured at three time points (baseline, 3-month, and 6-month post intervention).
  The PUMNS is a questionnaire used to assess neurological responses (reflexes) and spasticity in individuals with motor neuron disease (MND). It helps evaluate the severity of the disease and monitor changes in the patient's nervous system. The researcher will assess various reflexes and signs of spasticity, such as Hoffman's sign and Babinski's sign.
Patient health questionnaire (PHQ-9) | PHQ-9 will be measured at three time points (baseline, 3-month, and 6-month).
  The Patient Health Questionnaire-9 (PHQ-9) is a widely used self-report screening tool for assessing the presence and severity of depression. It consists of 9 items, each corresponding to one of the diagnostic criteria for major depressive disorder as defined by the DSM-IV. The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms.
EuroQol 5-Dimension 5-level (EQ-5D-5L) | EQ-5D-5L will be measure at three time ponts (baseline, 3-month, and 6-months post intervention).
  The EuroQol 5-Dimension 5-Level (EQ-5D-5L) is a standardized questionnaire used to measure health-related quality of life (HRQoL). It is widely used in clinical, public health, and economic evaluations to assess the overall health status of individuals. The EQ-5D-5L includes two parts: 1) Descriptive System whhich assesses health across five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and 2) EQ Visual Analogue Scale (EQ VAS - A vertical scale ranging from 0 (worst imaginable health) to 100 (best imaginable health) on which the respondent rates their overall health.
Forced vital capacity (FVC) | FVC will be measured at three time points (baseline, 3-month, and 6-month post intervention).
  Forced Vital Capacity (FVC) is a key measure of lung function that assesses the amount of air a person can forcefully exhale after taking the deepest possible breath. It is measured in litres (L) using a device called a spirometer.
  During the test, the person inhales fully and then exhales as hard and fast as possible until no more air can be expelled. The total volume of air exhaled is recorded as the FVC. This test helps evaluate lung capacity and is commonly used to monitor respiratory conditions such as asthma, chronic obstructive pulmonary disease (COPD), and motor neuron disease (MND).
Magnetic resonance imaging (MRI) | Brain imaging using MRI will be measured at three time points (baseline, 3-month and 6-month post intervention).
  Brain imaging using MRI is a technique used to measure cortical thickness by capturing high-resolution images of brain structures. Participants lie in an MRI scanner for approximately 10 to 20 minutes during data acquisition. After the scan, the images are processed using FreeSurfer software. Cortical thickness is calculated by measuring the distance between the white matter surface and the outer surface of the cerebral cortex.
Compound muscle action potential (CMAP) | CMAP will be meausred at three time points (baseline, 3-month, and 6-month post intervention).
  To record Compound Muscle Action Potential (CMAP), electrical stimulation is applied to the nerve, gradually increasing the intensity step by step. The muscle responses are recorded to determine the maximum CMAP response, which is achieved at supramaximal stimulation. CMAP is a key parameter in studies related to nerve conduction and provides important information about motor neuron function. A higher CMAP value indicates greater muscle fiber activation, which reflects the number of functional motor units still intact.

CONTACTS AND LOCATIONS:
Overall Officials: Jakkrit Amornvit, MD, Principal Investigator — Chulalongkorn University; Phunsuk Kantha, PT.,PhD, Principal Investigator — Mahidol University; Kulvara Lapanan, PT, Principal Investigator — Chulalongkorn University and Neuroscience Resesarch Australia
Locations (1):
- King Chulalongkorn Memorial hospital, The Thai Red Cross Society, Bangkok, Pathumwan, Thailand